CLINICAL TRIAL: NCT00377806
Title: A One Week, Double-Blind, Adaptive, Randomized, Multicenter Study to Compare the Efficacy, Safety and Tolerability of Topical Diclofenac Gel Versus Placebo in Patients With Superficial Thrombophlebitis
Brief Title: Topical Diclofenac Gel in Patients With Superficial Inflammation of the Veins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVOL458UDE01
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Superficial Thrombophlebitis of the Upper Limb
Keywords: Superficial thrombophlebitis, diclofenac gel, non steroidal antiinflammatory drugs

INTERVENTIONS:
Drug: Diclofenac gel

SUMMARY:
This study will assess the efficacy, safety and tolerability of topically administered diclofenac gel versus placebo with respect to the symptom score (pain, temperature and size of erythema along the superficial vein)

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of topical treatment for inflammatory, painful superficial thrombophlebitis of the upper limb
* Spontaneous or iatrogenic superficial thrombophebitis of the upper limb

Exclusion Criteria:

* Hypersensitivity to the study drug, to actylsalicyclic acid and other non-steroidal antirheumatic agents and to the ingredients of the gel
* Paitents who had developed asthma, skin reactions or acute rhinitis to acetylsalicylic acid or other non-steroidal antirheumatic agents in the past
* Therapy with varicose vein remedies, antithrombotic or antiphlogistic agents as well as corticosteroids for more than 7 days prior to study start
* Acute deep vein thrombosis and thrombophlebitis extending into other deep veins

Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The area under the curve (AUC) of the symptom score (pain, temperature and size of erythema along the superficial vein)

SECONDARY OUTCOMES:
Patient's global assessment of drug effect at each visit
Physician's global assessment of drug effect at each visit
AUC of assessment of pain (visual analog scale) between treatment day 1 and day 5
AUC of assessment of inflammatory area of the superficial thrombophlebitis between treatment day 1 and 5
AUC of assessment of temperature of inflammatory area around superficial thrombophlebitis between treatment day 1 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis, Nuremberg, Germany